CLINICAL TRIAL: NCT06669377
Title: Transcatheter Arterial Chemoembolization Combined With ICIs Plus MTT After Irradiation Stent Placement in HCC With Main PVTT: a Multicenter Propensity Score Matching Study
Brief Title: TACE Combined With ICIs Plus MTT After 125I Irradiation Stent Placement in HCC With Main PVTT.
Status: Recruiting | Type: Observational
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Prof., Zhongda Hospital
Other Study IDs: PATENCY2
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; irradiation stent; portal vein tumor thrombosis; immune checkpoint inhibitor; molecular targeted therapy; transcatheter arterial chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatocellular carcinoma (HCC) patients with Vp4 [main trunk] portal vein tumor thrombosis (PVTT) face a significantly poor prognosis, and current treatment options provide limited benefits. We aimed to assess the safety and efficacy of transcatheter arterial chemoembolization (TACE) combined with immune checkpoint inhibitors (ICIs) plus molecular targeted therapy (MTT) after irradiation stent placement (ISP) as first line treatment for HCC patients with Vp4 PVTT.

DETAILED DESCRIPTION:
According to the latest report, liver cancer is the third leading cause of cancer-related deaths, following lung and colorectal cancers, with hepatocellular carcinoma (HCC) accounting for 75% to 85% of all primary liver cancer cases. Portal vein tumor thrombosis (PVTT) is a significant indicator of poor prognosis in HCC, with a high incidence of 39-63% and a median survival of 2.7 months.

Systemic therapy is the recommended treatment for HCC patients with Vp4 [main trunk] portal vein tumor thrombus (PVTT). The landmark IMbrave150 study has ushered in a new era of combined systemic therapy for patients with unresectable HCC. However, subgroup analysis indicates that overall survival (OS) for HCC patients with Vp4 PVTT remains poor in both the sorafenib (5.5 months) or atezolizumab plus bevacizumab (7.6 months) groups.

Recent studies indicate that incorporating transcatheter arterial chemoembolization (TACE) significantly benefits HCC patients compared to systemic therapy alone, with significantly prolonged OS and progression free survival (PFS). However, HCC with PVTT is generally considered a contraindication to transcatheter arterial chemoembolization (TACE). When the portal vein blood supply has been damaged, TACE may lead to the reduction or even interruption of hepatic artery and the exacerbate the deterioration of liver function, eventually leading to liver failure. Although a few studies have explored TACE treatment in patients with Vp3-4 PVTT, the results have not shown a significant extension in survival.

Iodine-125 (125I) irradiation stent placement (ISP) can quickly restore blood flow and alleviate portal hypertension caused by tumor thrombus. Moreover, compared to bare stents, irradiation stents offer a uniform and sustained radiation distribution to PVTT, thus ensuring long-term patency of the portal vein and enabling the possibility of TACE for HCC patients with Vp4 PVTT. Our previous randomized controlled trial has demonstrated the safety and efficacy of ISP combined with TACE.

Herein, this nationwide multicenter, retrospective, propensity score matching (PSM) cohort study (PATENCYⅡ) aims to assess the safety and efficacy of immune checkpoint inhibitors (ICIs) plus molecular targeted therapy (MTT) with or without ISP plus TACE as first line treatment for HCC patients with Vp4 PVTT.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years old; (2) diagnosis of HCC is confirmed through histological or cytological analysis, as well as clinical features; (3) histologically confirmed or imaging-diagnosed PVTT extending to the main portal vein (Vp4); (4) including at least one measurable intrahepatic lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1; (5) Eastern Cooperative Oncology Group (ECOG) performance status of ≤2; (6) patients received first-line treatment with either ICIs-MTT or an ISP-containing quadruple combination within eight weeks (In the ICIs-MTT group, MTT was administered alongside ICIs. In the ISP-containing quadruple, TIT and ICIs-MTT were given after stent placement and portal vein recanalization, either simultaneously or within eight weeks before or after the ICIs-MTT therapy).

Exclusion Criteria:

1. patients with extrahepatic metastases; (2) a history of or concurrent malignancies; (3) patients underwent prior systemic treatments or locoregional therapies, including surgery, radiation therapy, hepatic arterial embolization, TACE, hepatic arterial infusion, radiofrequency ablation, percutaneous ethanol injection, and cryoablation, within three months before the initiation of ISP.; (4) Child-Pugh grade C liver function, a Child-Pugh score of 3 for ascites, or the presence of overt hepatic encephalopathy; (5) incomplete outcome data or missing essential baseline factors for analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HCC and Vp4 PVTT who received TACE in combination with PD-1/PD-L1 inhibitors and molecular target therapies after 125I irradiation stent placement under real-world practice conditions
Sampling Method: Probability Sample
Enrollment: 444 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 2 years
  The OS is defined as the time from the initiation of any combination treatment to death due to any cause.

SECONDARY OUTCOMES:
Progression free survival(PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | up to approximately 2 years
  The PFS is defined as the time from the initiation of any combination treatment to the first documented progressive disease (according to RECIST 1.1) or death due to any cause, whichever occurs first.
PFS per Modified Response Evaluation Criteria in Solid Tumors (mRECIST) | up to approximately 2 years
  The PFS is defined as the time from the initiation of any combination treatment to the first documented progressive disease (according to mRECIST) or death due to any cause, whichever occurs first.
Objective response rate(ORR) of intrahepatic lesions and portal vein tumor thrombosis (PVTT) per RESCIST 1.1 | up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented complete response(CR) or partial response(PR) per RECIST 1.1.
Objective response rate(ORR) of intrahepatic lesions and portal vein tumor thrombosis (PVTT) per mRECIST | up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented CR or PR per mRECIST.
Disease Control Rate (DCR) per RESCIST 1.1 | up to approximately 2 years
  DCR is defined as the percentage of participants who have a best overall response of CR, PR, or stable disease (SD)per RESCIST 1.1.
Disease Control Rate (DCR) per mRECIST | up to approximately 2 years
  DCR is defined as the percentage of participants who have a best overall response of CR, PR, or stable disease (SD) per mRECIST.
Adverse event(AE) per Common Terminology Criteria for Adverse Events(CTCAE) 5.0 | up to approximately 2 years
  The percentage and degree of patients who experience at least one AE, whether or not considered related to the treatment, according to CTCAE version 5.0.
Hepatic function | up to approximately 2 years
  Hepatic function was measured in terms of total bilirubin, albumin, aspartate transaminase, alanine aminotransferase, alkaline phosphatase, prothrombin time
Patency of portal vein | up to approximately 2 years
  Patency of portal vein was evaluated by color doppler ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Gaojun Teng, M.D., Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China